CLINICAL TRIAL: NCT06390943
Title: Low Birthweight and Preterm Infant Feeding Trial and Supportive Care Package (LIFT-UP): Implementation Research of an In-facility and Community Supportive Care Package in India, Malawi and Tanzania
Brief Title: Low Birthweight and Preterm Infant Feeding Trial and Supportive Care Package: Implementation Research
Acronym: LIFT-UP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Boston Children's Hospital (Other); Community Empowerment Lab (Other); Emory University (Other); Muhimbili University of Health and Allied Sciences (Other); Jawaharlal Nehru Medical College (Other); PATH (Other); University of North Carolina (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Katherine Semrau, Deputy Director, Ariadne Labs & Director, BetterBirth Program, Harvard School of Public Health (HSPH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB23-0273
Record Dates: First submitted 2024-03-30; First posted 2024-04-30 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-08

CONDITIONS: Low Birthweight; Preterm Birth
Keywords: Lactation support; Kangaroo Mother Care; WASH
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obj 1 Infants receiving facility-based FSP+; Obj 2 infants receiving transition-to-home FSP+ (Other)
  Interventions: Other: Facility-based feeding support package plus (FB-FSP+); Other: Transition-to-home feeding support package plus (TTH-FSP+)

INTERVENTIONS:
Other: Facility-based feeding support package plus (FB-FSP+) — Package of materials to support facility-based feeding and lactation, KMC and WASH, including a training curriculum, training guide, and implementation materials, such as Standard Operating Procedures (SOPs) and job aides
Other: Transition-to-home feeding support package plus (TTH-FSP+) — Package of materials to support transition-to-home feeding and lactation, KMC and WASH, including a training curriculum, training guide, and implementation materials, such as Standard Operating Procedures (SOPs) and job aides

SUMMARY:
Low Birthweight and Preterm Infant Feeding Trial and Supportive Care Package (LIFT-UP) aims to improve feeding and growth outcomes among low birthweight (LBW; <2.5kg) or preterm (<37 weeks gestational age) infants admitted to neonatal intensive care units (NICU) in India, Malawi, and Tanzania by (1) supporting the initiation, establishment, and maintenance of maternal lactation and prioritized provision of human milk, Kangaroo Mother Care (KMC) and appropriate water, sanitation and hygiene (WASH) practices; and (2) facilitating feeding counseling at home post-discharge from the facility.

DETAILED DESCRIPTION:
AIM: To improve feeding and growth outcomes among low birthweight (LBW; <2.5kg) or preterm (<37 weeks gestational age) infants admitted to NICUs in India, Malawi, and Tanzania by (1) supporting the initiation, establishment, and maintenance of maternal lactation and prioritized provision of human milk, Kangaroo Mother Care (KMC) and appropriate water, sanitation and hygiene (WASH) practices; and (2) facilitating feeding counseling at home post-discharge from the facility.

OBJECTIVES:

To implement and evaluate a co-designed facility-based lactation support/management and feeding counseling + KMC + WASH package (FB-FSP+: Facility-Based Feeding Support Package Plus) for LBW or preterm infants admitted to the neonatal intensive care unit (NICU) and their families from birth to discharge.

To implement and evaluate a co-designed, scalable transition-to-home lactation support/management and feeding counseling + KMC + WASH package (TTH-FSP+: Transition to Home Feeding Support Package Plus) for LBW or preterm infants discharged home from the NICU in India and their mothers/families.

STUDY DESIGN: This multi-site, mixed-methods adaptive implementation science research study will collect quantitative and qualitative data to evaluate the training of providers, the impact of each intervention on key infant feeding, growth, and other health outcomes, the feasibility and acceptability of each intervention for mothers and providers, and the overall experience of mother-infant dyads. Investigators will apply the RE-AIM framework to unpack Reach, Effectiveness, Adoption, Implementation, and Maintenance. Findings will lead to recommendations for iteration and scale-up of the FB- and TTH-FSP+. Investigators will evaluate multiple primary and secondary quantitative outcomes to assess effectiveness.

SAMPLE SIZE: Overall, investigators will enroll 695 participants, 50% in India, 50% in Malawi & Tanzania: up to 520 infants (463 mothers assuming 11% twin rate), 110 mothers (in-depth interviews), 30 healthcare providers, 15 study staff, and 20 community providers.

Objective 1: A sample of 80 infants and their mothers is sufficient to detect the effect sizes for each of the primary and secondary outcomes with 80% power, 0.05 alpha. Smaller improvements in key outcomes for the pre/post analysis can be detected for the implementation study (n=80 baseline vs 240 implementation) compared to the pilot study (n=80 baseline vs 80 pilot).

Objective 2: Investigators will conduct up to 40 in-depth interviews (IDIs) with providers and 20 with mothers. A sample of 60 infants and their mothers is sufficient to detect the effect sizes for each of the primary and secondary outcomes with 80% power, 0.05 alpha.

ENROLLMENT: OBJECTIVE 1 (FB-FSP+) Mother-infant dyads (quantitative): All infants born in a study facility will receive immediate maternal and newborn care per World Health Organization recommendations, including breast milk feeding/expression support within 1 hour. Inborn LBW or preterm infants admitted to the NICU will be screened for eligibility and their mothers consented.

Mothers (qualitative): Mothers will be recruited and consented before discharge from study facilities.

Research Nurses (qualitative): Research nurses providing the intervention will be consented prior to IDIs.

Healthcare providers (quantitative): Appropriate labor ward, NICU, and step-down ward providers will be identified by facility and NICU leadership/staff to implement the FB-FSP+ and consented.

Healthcare providers (qualitative): NICU providers will be recruited and consented during study implementation.

ENROLLMENT FOR OBJECTIVE 2 (TTH-FSP+, INDIA ONLY) Mothers (quantitative): Mothers exposed to Objective 1 will be recruited around the time of discharge and consented.

Community providers (quantitative): Community providers within a given cadre(s) who provide care to LBW or preterm infants within the catchment area will be recruited and consented.

Mothers (qualitative): Mothers receiving the TTH-FSP+ will be recruited and consented during study visits.

Community providers (qualitative): Community providers will be recruited and consented after beginning implementation of the TTH-FSP+.

STUDY INTERVENTION: The FB-FSP+ and the TTH-FSP+ will build on an existing Specialized Lactation Support and Newborn Nutrition for the Small and Sick Newborn Training curriculum to include support for KMC and WASH. The FSP+ will include a training guide, Standard Operating Procedures and job aids specific to each hospital's and community's needs identified through co-design workshops with key stakeholders that utilize human-centered design methods.

DATA COLLECTION FOR OBJECTIVE 1 (FB-FSP+) Data will be collected in 3 phases.

Baseline data collection will occur over 6 weeks among eligible mother-infant dyads prior to introducing the intervention. Baseline will be the comparison group for the implementation research study and the pilot study.

A 6-week pilot study conducted by research staff in each country will assess the acceptability, feasibility, and impact of the ideal delivery of the FB-FSP+. A quick final iteration of the FSP+ will occur before implementing in phase 3.

The FB-FSP+ will be implemented for 1 year using an adaptive models-based approach. Three consecutive models will be implemented for 4 months each. Investigators will collect panel data at 1.5, 5.5, and 10.5 months after the start of implementation for 1.5 months to assess effectiveness and inform model adaptations. Different mother-infant dyads will be surveyed at each time point to assess differences in the impact of implementation over time.

Prior to start, healthcare providers will be selected and trained to implement the FSP+ as part of their regular workload. They will complete a knowledge, attitudes, and practices (KAP) survey on lactation support/management, feeding, KMC, and WASH (1) prior to training, (2) immediately post-training, and (3) 6 months post-training.

Data collection with mother-infant dyads will take 1-2 hours at one time point between NICU admission and day of discharge during panel data collection. Mothers will be asked about their demographics, pregnancy history, health, and their infants' health. Study staff will take the mother's weight and height, the infants' weight, length, head circumference and mid-upper arm circumference (MUAC), and data from mothers' and infants' charts.

A subset of 60 mothers exposed to the FB-FSP+ will be interviewed by study staff, 30 of whom whose babies received care in the NICU within 1.5 months of implementation and another 30 whose babies received care within 5.5 months. Interviews will explore mothers' experiences and perceptions of the acceptability and feasibility of the FB-FSP+.

A subset of 15-30 healthcare providers across all sites will be interviewed per time point at 1.5 months and 5.5 months after implementing the FB-FSP+. Investigators aim to interview the same providers at both times to understand how implementation has affected their practices, skills and workload over time. Interviews will explore acceptability and feasibility of the FB-FSP+ and barriers and facilitators to its implementation.

DATA COLLECTION FOR OBJECTIVE 2 (TTH-FSP+, INDIA ONLY) Baseline data collection will occur before implementing the TTH-FSP+ among mothers exposed to the FB-FSP+ and discharged home. Data collection points will be on the day of discharge and at 2 and 6 weeks post-discharge.

The TTH-FSP+ will be implemented for 6 months, using an adaptive models-based approach. Three models will be consecutively implemented for 3 months each. Quantitative and qualitative analysis will begin after 2 months to inform model adaptations. Data collection points will be on the day of discharge and at 2 and 6 weeks post-discharge.

Community providers will be trained to deliver the TTH-FSP+ for dyads residing in a defined catchment area once they are discharged home. Community providers will complete a KAP survey on feeding counseling, KMC, and WASH at three timepoints: (1) just prior to training, (2) immediately post-training, and (3) 6 months post-training.

Data collection will begin on the day of discharge prior to leaving the facility, and mothers will respond to questions about their demographics, pregnancy history, health, and their infants' health. During 2 home visits, mothers will respond to questions on breastfeeding self-efficacy and health, as well as their infants' health and feeding practices. Mothers' weight and height will be measured at one study visit. The infants' weight, length, head circumference and MUAC will be measured at each study visit.

Interviews with mothers will be done at 6 weeks post-discharge during implementation of Model 1 & 2 and will explore their experiences with the TTH-FSP+ and their perspectives on its acceptability and feasibility .

Interviews with community providers will be conducted once during implementation of each Model 1 & 2. Investigators aim to interview the same providers at both time points. Interviews will explore community providers' experiences delivering the TTH-FSP+ and their perspectives on its acceptability and feasibility.

ELIGIBILITY:
OBJECTIVE 1 (FACILITY-BASED)

Inclusion criteria

Infants

* Low birthweight (≤2.5kg) or preterm (<37 weeks) infants admitted to NICU at study facility
* In-born infants admitted to the NICU within 24 hours of birth)
* Mother and infant alive during screening
* Mother consents for herself and infant
* Women (mothers) who are age of majority: Tanzania and India: 18+; Malawi: 16-17 and married OR 18+

Healthcare providers

* Healthcare provider who was trained to deliver the facility-based FSP+
* Healthcare provider consents for him/herself

Exclusion criteria

Infants

* Out-born infants referred to study facility NICU
* Congenital anomalies or acquired conditions that interfere with feeding or placement of nasogastric/ orogastric (NG/OG) tube [e.g., cleft lip/palate, toxoplasmosis,other agents, rubella, cytomegalovirus, and herpes (TORCH), Trisomy 21, Congenital cardiac defect, neural tube defect, gastrointestinal (GI) tract anomalies, hydrocephalus, necrotizing enterocolitis]
* Severe birth asphyxia
* Unknown date of birth and unknown gestational age

OBJECTIVE 2 (TRANSITION-TO-HOME)

Inclusion criteria

Infants

* Infants in India-Uttar Pradesh site
* LBW (<2.5kg) or preterm (<37 weeks) infants discharged from a study facility and fulfilling all objective 1 inclusion criteria (exposed to objective 1 intervention)
* Lives within catchment areas of study facility (50km)
* Mother intends to stay in the catchment areas for 3 months post-birth with infant

Community providers

* Community provider who was trained to deliver the transition-to-home FSP+.
* Community provider consents for him/herself

Exclusion criteria

Infants

* Not screened and was not exposed to objective 1 intervention (and meet all eligibility criteria)
* Lives outside the defined catchment area
* Mother does not intend to stay in the catchment areas for 3 months post-birth with infant

Community providers

-Community provider who was not trained to deliver the transition-to-home FSP+.

Min Age: 1 Minute | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 695 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Obj 1: Early initiation of mother's breast milk feeding | 1 hour after birth
  % infants initiated breast milk feeding within 1 hour of birth
Obj 1: Early initiation of mother's first breast stimulation | 1 hour after birth
  % mothers initiated breast stimulation via first breast milk expression or baby first put to breast within 1 hour of birth
Obj 1: Number of sessions when infant was fed mother's direct or expressed breast milk in previous 24 hours | 24 hours
  Mean number of mother's breast milk feeding sessions (direct or expressed) in the last 24 hours
Obj 1: Number of mother's breast milk expression sessions in previous 24 hours | 24 hours
  Mean number of sessions in which mother expressed breast milk in the last 24 hours
Obj 1 & 2: Maternal breastfeeding self-efficacy/confidence | Obj 1 Pilot: On day of facility discharge or at 2 weeks age (whichever is first); Obj 1 Implementation: 1.5, 5.5 and 10.5 months after the start of study implementation; Obj 2: On day of enrollment and 2 weeks and 6 weeks later
  Mean score (range 14-70) on validated Breastfeeding Self-Efficacy Scale-Short Form; higher scores reflect more significant levels of breastfeeding self-efficacy
Obj 2: Growth velocity (g/kg/d) | 6 weeks after initial facility discharge
  Mean change in infant's weight (growth) calculated in grams/kilogram/day (g/kg/ day) from facility discharge to study discharge

SECONDARY OUTCOMES:
Obj 1: Time of first feed of mother's breast milk in NICU | From date/time of enrollment until date/time of first documented feed on mother's breast milk in the NICU, assessed up to facility discharge or 14 days, whichever comes first
  Mean time from NICU admission to first feed of mother's breast milk in NICU
Obj 1: Growth velocity (g/kg/d) | Obj 1 Pilot: Birth to day of discharge or 2 weeks of age (whichever is first); Obj 1 Implementation: 1.5, 5.5 and 10.5 months after the start of study implementation
  Mean change in infant's weight (growth) calculated in grams/kilogram/day (g/kg/ day) from birth to facility discharge
Obj 1: 20g/kg/day weight gain | Obj 1 Pilot: Birth to facility discharge or 2 weeks of age; Obj 1 Implementation: 1.5, 5.5 and 10.5 months after the start of study implementation
  Obj 1 Pilot: % infants who experienced a change in weight of at least 20g/kg/day between birth and day of discharge or 2 weeks of age; Obj 1 Implementation: % infants who experienced a change in weight of at least 20g/kg/day between birth and day of evaluation (varies by infant)
Obj 1 & 2: Infants fed exclusively on mother's own milk in the previous 24 hours | 24 hours
  % infants fed exclusively mother's own milk in the last 24 hours
Obj 1 & 2: Infants receiving KMC in previous 24 hours | 24 hours
  % infants receiving any Kangaroo Mother Care in the last 24 hours
Obj 1 & 2: Infants receiving at least 8 hours of KMC in last 24 hours | 24 hours
  % infants receiving at least 8 hours of Kangaroo Mother Care in last 24 hours
Obj 1 & 2: Management of feeding difficulties | Obj 1 Pilot: Daily referring to the 24 hours assessed from enrollment until facility discharge or 2 weeks of age (whichever occurs first); Obj 1 Implementation: 1.5, 5.5 and 10.5 months after the start of study implementation
  % of feeding difficulties that mothers reported which were resolved through support
Obj 2: Number of sessions when infant was fed mother's direct or expressed breast milk in previous 24 hours | 24 hours
  Mean number of mother's breast milk feeding sessions (direct or expressed) in the last 24 hours
Obj 2: Number of mother's breast milk expression sessions in previous 24 hours | 24 hours
  Mean number of sessions in which mother expressed breast milk in the last 24 hours

OTHER OUTCOMES:
Obj 1 & 2: % infants who receive the "minimum package" | Obj 1 Pilot: At discharge or at 2 weeks age (whichever is first); Obj 1 Implementation: 1.5, 5.5 and 10.5 months after the start of study implementation; Obj 2: On day of enrollment and 2 weeks and 6 weeks later
  The minimum package will be defined and likely be based on milestones that vary by length of stay and perhaps baby status
Obj 1: Feeding competency | Difference between enrollment (within 24 hours of birth) and day of discharge or 2 weeks of age (whichever is first)
  Pilot only: Mean feeding competency score on on Preterm Infant Breastfeeding Behavior Scale (range 0-20); % of mother-infant dyads who score >15 on Preterm Infant Breastfeeding Behavior Scale; Mature breastfeeding behavior is indicated if the newborn achieves the highest scores on all six items.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Semrau, PhD, MPH, Principal Investigator — Ariadne Labs
Locations (5):
- India (3):
  - Ganesh Shankar Vidyarthi Memorial Medical College, Kanpur
  - King George Medical College, Lucknow
  - Institute of Medical Sciences, Banaras Hindu University, Varanasi
- Bwaila District Hospital, Lilongwe, Malawi
- Amana Regional Hospital, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets will be released after the close of the project in a data sharing repository, such as Harvard Dataverse or similar, in a format readable by analytics tools. Harvard Dataverse is an online data repository where you can share, preserve, cite, explore, and analyze research data. Data sets and data dictionaries will be provided in compliance with the ethical review boards' requirements. As part of the Harvard Dataverse system, registration to download datasets is required. External partners (those not involved in the study) must provide their contact information and describe their intention of data use.
Supporting Information: Study Protocol, SAP, CSR